CLINICAL TRIAL: NCT03920137
Title: Adaptation and Initial Evaluation of Transdiagnostic CBT for Anxious and Depressed Smokers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Michael J. Zvolensky, Ph.D., Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000859
Record Dates: First submitted 2018-04-18; First posted 2019-04-18 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Standard of Care; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active- UP-ST (Active Comparator): The intervention will be the UP-ST therapy sessions. Treatment will be delivered using the new UP-ST protocol that will be developed in Phase I by integrating components of smoking cessation treatments (e.g. using the nicotine patch) with the theoretical model and treatment components of the existing UP treatment protocol, which includes both a therapist14 and patient12 manual. The UP-ST will maintain the same focus on transdiagnostic mechanisms of change as in the original UP, but will be adapted to integrate the smoking cessation focus and concurrent use of NRT. Thus, the investigators can successfully adapt and develop the new UP-ST to be delivered in eight 90-minute sessions and will be able to incorporate content from each of the 8 modules of the UP in the new UP-ST protocol.
  Interventions: Behavioral: UP-ST Therapy; Device: Nicotine Patch
- Control- Standard (Experimental): The Intervention will be the standard therapy sessions. Participants will receive a standard smoking cessation treatment based on the most recent clinical practice guideline from the U.S. Department of Health and Human Services, Treating Tobacco Use and Dependence19. The investigative team has considerable expertise in developing and evaluating behavioral and pharmacological treatments for smoking cessation. Treatment will be delivered in eight, 90-minute sessions over an eight-week period.
  Interventions: Behavioral: Standard Therapy

INTERVENTIONS:
Behavioral: UP-ST Therapy — Phase 1 analyses will focus primarily on demonstrating feasibility and utility of the new UP-ST intervention. Feasibility will be determined by examining the proportion of individuals who 1) complete each module of the UP-ST treatment, 2) complete a full course of the UP-ST treatment, and by 3) benchmarking participant ratings of treatment credibility, expectancy, and satisfaction with corresponding ratings from our previous clinical trials examining the UP or ST interventions. The investigators will include and examine outcomes on the same measures that will be used in phase 2, but due to the sample size our analyses for Phase 1 will focus on intraindividual effect sizes (with 95% CI) for continuous smoking, anxiety, and depression outcomes
  Arms: Active- UP-ST
Behavioral: Standard Therapy — In the control group therapists will hold standard smoking cessation therapy sessions.
  Arms: Control- Standard
Device: Nicotine Patch — Nicotine patches will be worn in tandem with UP-ST therapy
  Arms: Active- UP-ST

SUMMARY:
This study will look at the effectiveness of a new treatment protocol for anxious and depressed smokers. Participants with clinically significant anxiety or depression will receive either the standard smoking cessation treatment or the Unified Protocol for Smoking Cessation Treatment. This study will demonstrate that a single treatment protocol can effectively address both smoking and the complex emotional comorbidities that are widespread in smokers will provide a novel, impactful, and highly disseminable treatment option missing from today's smoking cessation arsenal.

DETAILED DESCRIPTION:
The present proposal aims to develop a new and efficient treatment for smokers with clinically significant anxiety or depression. In Phase I, the investigators will complete the development of a new treatment protocol (Unified Protocol for Smoking Cessation Treatment; UP-ST) that integrates current best practices of cognitive behavioral smoking cessation treatments and nicotine replacement therapy with the recently developed UP treatment protocol that has been shown to effectively treat both anxiety disorders and depression and to impact specific mechanisms (e.g., neuroticism) that are relevant to both smoking and anxiety/depression remission. In Phase II, 60 smokers with clinically significant anxiety or depression will be recruited and randomly assigned to either: (1) the UP-ST or (2) standard smoking cessation treatment (ST) based on the most recent clinical practice guideline from the U.S. Department of Health and Human Services. The investigators will examine the UP-ST relative to ST on smoking, anxiety/depression, and mechanisms of change. Demonstrating that a single treatment protocol can effectively address both smoking and the complex emotional comorbidities that are widespread in smokers will provide a novel, impactful, and highly disseminable treatment option missing from today's smoking cessation arsenal.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion criteria for the study include 1) being 18-65 years of age, 2) daily smoking of at least 5 cigarettes per day for at least one year and biochemically confirmed at least 10 ppm at baseline. Participants must be 3) motivated to quit smoking in the next month 4) have clinically significant anxiety or depression defined as >=8 on the OASIS or ODIS, 5) must be willing and able to attend all the appointments, and 6) must be willing to quit smoking as the sixth treatment session.

Exclusion Criteria:

- Exclusion criteria include 1) Use of other tobacco products 2) Report of current or intended participation in a concurrent substance abuse treatment, 3) Ongoing psychotherapy of any duration targeting anxiety or depression, 4) Current non-nicotine substance dependence, 5) Not being fluent in English, 6) Current use of any pharmacotherapy or psychotherapy for smoking cessation not provided by the researchers, 7) Legal status that will interfere with participation, 8) Positive pregnancy test at baseline, 9) Active suicidality (i.e., suicidal ideation, intent, and/or plan) or current psychosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-12-20 (Actual); Primary Completion 2023-07-26 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Short- and long-term point prevalence abstinence (PPA). | 12 months
  In three separate follow up appointments, one 3 months after the end of treatments, one 6 months after and one 12 months after, The investigators will ask participants various questions about their abstinence. The investigators will measure the length of time between when treatment ends and when/ if they start smoking again. The unit of measure will be length of time in days. The investigators expect that point prevalence abstinence will be higher, both in the short term and long term, in the UP-ST condition than in the ST condition. Similarly, The investigators expect the rate of decline in abstinence over time to be shallower (smaller) in UP-ST than in ST.

SECONDARY OUTCOMES:
Tobacco withdrawal | 12 months
  In three separate follow up appointments 3, 6 and 12 months after the end of treatment, The investigators will administer a survey to participants. The survey will assess withdrawal symptoms. Participants will score this condition on a scale from 0-10. 10 meaning extremely severe and 0 meaning not at all. The investigators expect the mean score to be higher in the ST condition than the UP-ST condition at all time points.
Time to first smoking lapse and time to relapse | 12 months
  The investigators will ask participants to record the time (in days) of their first (if any) lapse in smoking and their relapse. The investigators will take an average for control and active participants and The investigators expect mean time to first lapse and to relapse to be greater for those in the UP-ST compared to those in the ST condition.
Tobacco craving | 12 months
  In three separate follow up appointments 3, 6 and 12 months after the end of treatment, The investigators will administer a survey to participants. The survey will assess tobacco craving. Participants will score this condition on a scale from 0-10. 10 meaning extremely severe and 0 meaning not at all. The investigators expect the mean score to be higher in the ST condition than the UP-ST condition at all time points.
Tobacco dependence | 12 months
  In three separate follow up appointments 3, 6 and 12 months after the end of treatment, The investigators will administer a survey to participants. The survey will assess tobacco dependence. Participants will score this condition on a scale from 0-10. 10 meaning extremely severe and 0 meaning not at all. The investigators expect the mean score to be higher in the ST condition than the UP-ST condition at all time points.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zvolensky, Ph.D., Principal Investigator — University of Houston; Matthew Gallagher, Ph.D., Study Director — University of Houston
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Data will be made available upon request.

REFERENCES:
- [Background] Zvolensky MJ, Jardin C, Wall MM, Gbedemah M, Hasin D, Shankman SA, Gallagher MW, Bakhshaie J, Goodwin RD. Psychological Distress Among Smokers in the United States: 2008-2014. Nicotine Tob Res. 2018 May 3;20(6):707-713. doi: 10.1093/ntr/ntx099. PMID 28482108
- [Background] National Center for Chronic Disease Prevention and Health Promotion (US) Office on Smoking and Health. The Health Consequences of Smoking-50 Years of Progress: A Report of the Surgeon General. Atlanta (GA): Centers for Disease Control and Prevention (US); 2014. Available from http://www.ncbi.nlm.nih.gov/books/NBK179276/ PMID 24455788